CLINICAL TRIAL: NCT06511245
Title: WEB™ Embolization System in the Treatment of Acutely Ruptured Intracranial Aneurysms Versus Other Endovascular Techniques
Brief Title: European, Multi-center, Exploratory Trial to Assess WEB Versus Other Endovascular Treatment in Ruptured Aneurysms.
Acronym: WAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP EMEA 23-01; CIP EMEA 23-01 (Other: Sponsor ID)
Record Dates: First submitted 2024-06-26; First posted 2024-07-19 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Ruptured Aneurysm
MeSH Terms: conditions — Aneurysm, Ruptured

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WEB (Other)
  Interventions: Other: Randomisation
- Other endovascular techniques (Other)
  Interventions: Other: Randomisation

INTERVENTIONS:
Other: Randomisation — Technique assigned through randomization

SUMMARY:
Comparison of efficacy and safety between WEB and other endovascular techniques

ELIGIBILITY:
Main Inclusion Criteria:

* Patient is above 18 years of age at the time of consent
* Patient has an identified acutely ruptured intracranial aneurysm requiring endovascular treatment (for the purposes of this study an acutely ruptured IA patient is defined as a patient with computed tomography (CT), magnetic resonance imaging (MRI), or lumbar puncture (LP) evidence of subarachnoid hemorrhage attributed to the index aneurysm within the last 30 days)
* Aneurysm dome diameter must be ≤ 10mm and within the diameter (and parent vessel diameter, as appropriate) range treatable by commercially available WEB devices as well as at least one other alternative commercially available endovascular treatment device used per hospital standard practice
* Aneurysm is located on the anterior communicating artery complex segment (ACom), internal carotid artery terminus (ICAt), anterior cerebral artery (ACA), middle cerebral artery (MCA), basilar apex, posterior communicating artery (PCom) or pericallosal artery
* Patient must be neurologically stable with a Hunt & Hess score of I to III
* Patient or patient's legally authorized representative (LAR) has provided written informed consent

Main Exclusion Criteria:

* Aneurysm to be treated is unsuitable for endovascular treatment with commercially available WEB devices and/or all other available endovascular treatment techniques used per standard site practice
* Patient presenting as target aneurysm a blister like or dissecting aneurysm
* Patient has more than one aneurysm requiring treatment within 30 days of completion of treatment of the target aneurysm
* Patient with multiple aneurysms in whom ruptured aneurysm cannot be identified
* Patient has pre-morbid mRS > 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
As exploratory design, one of the outcome will be the assessment of aneurysm occlusion at 12 months using Raymond-Roy scale. | 12 months (-3/+6 months)
  Raymond-Roy Classification is an angiographic classification including 3 classes, from class 1 (complete obliteration) to class 3 (aneurysm remnant).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Reims, Reims, France